CLINICAL TRIAL: NCT05094102
Title: Intraoperative Evaluation of Axillary Lymphatics for Breast Cancer Patients Undergoing Axillary Surgery
Brief Title: Intraoperative Evaluation of Axillary Lymphatics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institutes of Health (NIH) (NIH); OnLume Inc. (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW20058; 2020-0939 (Other: Institutional Review Board); A539713 (Other: UW Madison); SMPH/SURGERY/SURG ONC (Other: UW Madison); Protocol Version 11/3/2022 (Other: UW Madison); 2R44CA206754-02A1 (NIH)
Record Dates: First submitted 2021-09-08; First posted 2021-10-26 (Actual); Results first posted 2024-05-23 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-10

CONDITIONS: Lymphedema; Surgery; Breast Cancer
MeSH Terms: conditions — Lymphedema; Breast Neoplasms | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Axillary Surgery (Experimental): Breast cancer patients undergoing SLN biopsy (n=0-20) or axillary lymph node dissection (n=0-15) will be enrolled to undergo standard of care axillary reverse mapping (ARM) using isosulfan blue dye. Participants will also receive ICG injection with visualization through the OnLume Imaging System to allow comparison of blue dye versus ICG lymphatic identification.
  Interventions: Device: OnLume Imaging System; Drug: Indocyanine green

INTERVENTIONS:
Device: OnLume Imaging System — for fluorescence-guided surgery with ICG dye
Drug: Indocyanine green — Indocyanine green is a cyanine dye used in medical diagnostics
  Other Names: ICG

SUMMARY:
This study will assess the feasibility of using the OnLume Imaging System for fluorescence-guided surgery along with indocyanine green (ICG) dye in the operating room for the axillary reverse mapping (ARM) procedure in women with breast cancer scheduled to have axillary dissection (AD) or sentinel lymph node (SLN) biopsy.

DETAILED DESCRIPTION:
Lymphatic drainage from the upper arm is often different from that of the breast, allowing safe removal of only the lymphatics of the breast and protection of the lymphatic channels draining the upper extremity during axillary dissection (AD) or sentinel lymph node (SLN) biopsy, thereby reducing the risk of arm lymphedema.

In this prospective study, breast cancer patients undergoing SLN biopsy (n=0-20) or axillary lymph node dissection (n=0-15) will be enrolled to undergo axillary reverse mapping (ARM) using isosulfan blue dye. Participants will also receive ICG injection with visualization through the OnLume Imaging System to allow comparison of blue dye versus ICG lymphatic identification.

The standard of care (blue dye) will be used for clinical care while the OnLume Imaging System is being used to determine feasibility of the product.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Diagnosis of breast cancer requiring surgical lymph node evaluation either by sentinel lymph node biopsy or axillary lymph node dissection
* Surgery at University of Wisconsin Hospital and Clinic

Exclusion Criteria:

* Pregnant or breast feeding
* Unable to provide informed consent
* Allergy to indocyanine green
* Patients with clinically positive lymph nodes undergoing sentinel lymph node biopsy, with or without axillary lymph node dissection, after neoadjuvant chemotherapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2023-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather B Neuman, MD, MS, FACS, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at UW Hospital and Clinics from May 2022 to April 2023.
Period: Overall Study
Arm/Group | Axillary Surgery
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Axillary Surgery
Number analyzed (Participants) | 9
Age, Customized [Count of Participants; unit: Participants]
  30 to 39 years old | 1
  40 to 49 years old | 0
  50 to 59 years old | 3
  60 to 69 years old | 1
  70 to 79 years old | 3
  80 to 89 years old | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Cases Where Lymphatics Were Visualized by Blue Dye Versus by ICG Using the OnLume Imaging System
Description: This measure will determine whether lymphatics were visualized (yes/no) by each modality during axillary reverse mapping
Time Frame: up to 1 day (day of surgery)
Measure: Count of Participants; unit: Participants
Arm/Group | Axillary Surgery
Number analyzed (Participants) | 9
Participants
  Visualized by Blue Dye | 5
  Visualized by ICG | 9

2. Primary Outcome: Number of Cases Where Lymphatics Were Spared by Blue Dye Versus by ICG Using the OnLume Imaging System
Description: This measure will determine whether lymphatics were spared (yes/no) by each modality during axillary reverse mapping
Time Frame: up to 1 day (day of surgery)
Measure: Count of Participants; unit: Participants
Arm/Group | Axillary Surgery
Number analyzed (Participants) | 9
Participants
  Lymphatics spared by blue dye | 1
  Lymphatics spared by ICG | 5

3. Secondary Outcome: Maximum Contrast-to-Noise Ratio of ICG/OnLume Imaging System Fluorescence Signal
Description: A time curve of contrast-to-noise (CNR) ratio of lymphatic vessels to background tissue will be measured over the time frame of up to five minutes post-injection. The fluorescence signal intensity in both (1) the lymphatic vessels and in (2) the surrounding tissue will be measured in fluorescence arbitrary units. These two values will be aggregated to calculate and report the CNR, which is a unitless ratio. The maximum CNR will be reported.
Time Frame: Imaging data will be collected on the day of surgery (Day 1) - CNR will be measured up to five minutes post-injection of ICG]
Measure: Mean (Inter-Quartile Range); unit: Maximum CNR Ratio
Arm/Group | Axillary Surgery
Number analyzed (Participants) | 9
Maximum CNR Ratio | 54.9 [16.7 to 35.0]

ADVERSE EVENTS:
Time Frame: up to 1 day (day of surgery)
Arm/Group | Axillary Surgery
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-03): https://cdn.clinicaltrials.gov/large-docs/02/NCT05094102/Prot_SAP_001.pdf
  • Informed Consent Form (2022-12-05): https://cdn.clinicaltrials.gov/large-docs/02/NCT05094102/ICF_000.pdf